CLINICAL TRIAL: NCT04377035
Title: The ECHOVID-19 Study - A Prospective Cohort Study Investigating the Acute Effect of COVID-19 on the Heart and Lung by Ultrasound
Brief Title: The Role of Ultrasound in COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Tor Biering-Sørensen, Associate professor and Research Director, Cardiovascular Non-Invasive Imaging Research Laboratory, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-20021500
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective clinical cohort study of consecutive patients hospitalized at all hospitals of greater Copenhagen with a laboratory confirmed diagnosis of COVID-19. The investigators aim to examine if echocardiography - both conventional and advanced - can be used to predict which patients will develop acute respiratory distress syndrome (ARDS) or other short-term acute complications, especially focusing on cardiovascular outcomes. In addition, using a novel technique of lung ultrasound (LUS), The investigators aim to analyze specific LUS-findings, and associate them with short-term prognosis and development of ARDS and long-term cardiovascular morbidity and mortality. In all patients included, The investigators aim to examine long-term complications at timepoints: 2, 5 and 10 years of follow-up and examine if echocardiography - alone and in combination with biomarkers - can be used to detect early signs of cardiac complications and predict long-term risk of cardiovascular morbidity and mortality following COVID-19 infection

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized at hospitals of greater Copenhagen area and Zealand with a laboratory confirmed diagnosis of COVID-19 > 18 years of age.

Exclusion Criteria:

* Persons not able to cooperate
* Persons unable to understand and sign "informed consent"

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In.patients from hospitals of the greater Copenhagen area
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality during hospitalization and a confirmed COVID-19 diagnosis | 2.5 months
Incident ARDS (Adult Respiratory Distress Syndrome) and intensive care unit admission during hospitalization and a confirmed COVID-19 diagnosis | 2.5 months
Incident hypoxic respiratory failure during hospitalization and a confirmed COVID-19 diagnosis | 2.5 months

SECONDARY OUTCOMES:
Incident pulmonary embolism during hospitalization and a confirmed COVID-19 diagnosis | 2.5 months
Incident cardiac arrest during hospitalization and a confirmed COVID-19 diagnosis | 2.5 months
Death from any cause after hospital admission with a confirmed COVID-19 diagnosis at follow-up | 2.5 months to 10 years
Incident stroke after hospital admission with a confirmed COVID-19 diagnosis at follow-up | 2.5 months to 10 years
Incident heart failure after hospital admission with a confirmed COVID-19 diagnosis at follow-up | 2.5 months to 10 years
Incident myocardial infarction after hospital admission with a confirmed COVID-19 diagnosis at follow-up | 2.5 months to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, PhD, MPH, Principal Investigator — Research Director
Locations (1):
- Cardiovascular Non-Invasive Imaging Research Laboratory, department of Cardiology, Herlev & Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wodschow HZ, Davidovski FS, Christensen J, Lassen MCH, Skaarup KG, Nygaard H, Moller N, Rungby J, Biering-Sorensen T, Rossing P, Jensen NJ, Laursen JC. Oral ketone esters acutely improve myocardial contractility in post-hospitalized COVID-19 patients: A randomized placebo-controlled double-blind crossover study. Front Nutr. 2023 Feb 9;10:1131192. doi: 10.3389/fnut.2023.1131192. eCollection 2023. PMID 36845050
- [Derived] Olsen FJ, Lassen MCH, Skaarup KG, Christensen J, Davidovski FS, Alhakak AS, Sengelov M, Nielsen AB, Johansen ND, Graff C, Bundgaard H, Hassager C, Jabbari R, Carlsen J, Kirk O, Lindholm MG, Wiese L, Kristiansen OP, Nielsen OW, Lindegaard B, Tonder N, Ulrik CS, Lamberts M, Sivapalan P, Gislason G, Iversen K, Jensen JUS, Schou M, Svendsen JH, Aalen JM, Smiseth OA, Remme EW, Biering-Sorensen T. Myocardial Work in Patients Hospitalized With COVID-19: Relation to Biomarkers, COVID-19 Severity, and All-Cause Mortality. J Am Heart Assoc. 2022 Oct 4;11(19):e026571. doi: 10.1161/JAHA.122.026571. Epub 2022 Sep 21. PMID 36129046
- [Derived] Espersen C, Platz E, Alhakak AS, Sengelov M, Simonsen JO, Johansen ND, Davidovski FS, Christensen J, Bundgaard H, Hassager C, Jabbari R, Carlsen J, Kirk O, Lindholm MG, Kristiansen OP, Nielsen OW, Jeschke KN, Ulrik CS, Sivapalan P, Iversen K, Staehr Jensen JU, Schou M, Skaarup SH, Hojbjerg Lassen MC, Skaarup KG, Biering-Sorensen T. Lung ultrasound findings following COVID-19 hospitalization: A prospective longitudinal cohort study. Respir Med. 2022 Jun;197:106826. doi: 10.1016/j.rmed.2022.106826. Epub 2022 Apr 2. PMID 35453059
- [Derived] Espersen C, Platz E, Skaarup KG, Lassen MCH, Lind JN, Johansen ND, Sengelov M, Alhakak AS, Nielsen AB, Bundgaard H, Hassager C, Jabbari R, Carlsen J, Kirk O, Lindholm MG, Kristiansen OP, Nielsen OW, Jeschke KN, Ulrik CS, Sivapalan P, Gislason G, Iversen K, Jensen JUS, Schou M, Skaarup SH, Biering-Sorensen T. Lung Ultrasound Findings Associated With COVID-19 ARDS, ICU Admission, and All-Cause Mortality. Respir Care. 2022 Jan;67(1):66-75. doi: 10.4187/respcare.09108. Epub 2021 Nov 23. PMID 34815326
- [Derived] Skaarup KG, Lassen MCH, Espersen C, Lind JN, Johansen ND, Sengelov M, Alhakak AS, Nielsen AB, Ravnkilde K, Hauser R, Schops LB, Holt E, Bundgaard H, Hassager C, Jabbari R, Carlsen J, Kirk O, Bodtger U, Lindholm MG, Wiese L, Kristiansen OP, Walsted ES, Nielsen OW, Lindegaard B, Tonder N, Jeschke KN, Ulrik CS, Lamberts M, Sivapalan P, Pallisgaard J, Gislason G, Iversen K, Jensen JUS, Schou M, Skaarup SH, Platz E, Biering-Sorensen T. Lung ultrasound findings in hospitalized COVID-19 patients in relation to venous thromboembolic events: the ECHOVID-19 study. J Ultrasound. 2022 Sep;25(3):457-467. doi: 10.1007/s40477-021-00605-8. Epub 2021 Jul 2. PMID 34213740